CLINICAL TRIAL: NCT03913429
Title: Effects of Ultrasound-guided Bilateral Suprazygomatic Maxillary Nerve Block on Postoperative Pain After Elective Bimaxillary Osteotomy in Adult Patients
Brief Title: Ultrasound-guided Bilateral Suprazygomatic Maxillary Nerve Block and Bimaxillary Osteotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Servei Central d'Anestesiologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCAnestalia
Record Dates: First submitted 2019-03-11; First posted 2019-04-12 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Dentofacial Deformities; Regional Anesthesia Morbidity
Keywords: Orthognathic Surgery; Maxillary nerve blockade
MeSH Terms: conditions — Dentofacial Deformities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Infiltration performed by the surgeon at the intraoral and intranasal submucosal level in the maxilla (blockage of terminal branches of the maxillary nerve) after intubation and previous to surgical incision.
  A total of 50ml of the following preincisional mixture is infiltrated: ½ amp Adrenaline + 1amp Lidocaine 2% in physiological saline (SF) 100ml.
  Interventions: Procedure: Infiltration
- Study Group (Experimental): Bilateral ultrasound-guided maxillary nerve block by suprazygomatic route after intubation and previous to surgical incision performed by the anesthesiologist.
  A total of 5ml of Ropivacaine 0.37% infiltrated on each side.
  Interventions: Procedure: Maxillary nerve blockade

INTERVENTIONS:
Procedure: Infiltration — Infiltration performed by the surgeon at the intraoral and intranasal submucosal level in the maxilla (blockage of terminal branches of the maxillary nerve) after intubation and previous to surgical incision.
  A total of 50ml of the following preincisional mixture is infiltrated: ½ amp Adrenaline + 1amp Lidocaine 2% in physiological saline (SF) 100ml
  Other Names: Infiltration in the maxilla
  Arms: Control Group
Procedure: Maxillary nerve blockade — Bilateral ultrasound-guided maxillary nerve block by suprazygomatic route after intubation and previous to surgical incision performed by the anesthesiologist.
  A total of 5ml of Ropivacaine 0.37% infiltrated on each side. Together with adrenaline infiltration performed by the surgeon at the intraoral and intranasal submucosal level in the maxilla.
  A total of 50ml of the following preincisional mixture is infiltrated: ½ amp Adrenaline + 110ml SF.
  Other Names: Ultrasound guided Maxillary nerve blockade
  Arms: Study Group

SUMMARY:
Bimaxillary osteotomy is a surgery procedure of the orthognathic surgery field with the aim to correct dental and facial abnormalities, for both functional and aesthetic cases. The incidence of this abnormality is 5-10% of the population, and its etiology is unknown, with genetic, environmental and embryonic factors related. The surgical technique is complex, and requires osteotomy of the maxillary and jaw, which allows toward, forward, impact and rotation of these bones to fix the edges of the face. The anesthetic management of these patients is a challenge because of the difficult airway management and the perioperative pain control. Multimodal approach for pain control is a fact, and the use of local and regional anesthesia is mandatory. The investigators propose bilateral suprazygomatic maxillary nerve block for a proper control of postoperative pain after bimaxillary osteotomy.

DETAILED DESCRIPTION:
Bimaxillary osteotomy is a surgical procedure in the field of orthognathic surgery (from Latin, "ortho" straight and "gnatho" jaw) for the correction of dentofacial deformities, both for functional and aesthetic reasons. The incidence of this deformity is estimated to be around the 5-10% of the population. Genetic, environmental and embryonic factors are postulated to be the origin of such deformity, though its origin is still unknown. The surgical technique is complex, with the performance of mandibular and upper jaw osteotomies that allow to advance, retrude, impact and rotate these bones, to align the facial axes. For all these reasons, the anesthetic management of these patients is a challenge. First, the foreseeable difficulty of managing the patient's airway; and second, the control of the patient's pain in the perioperative period.

Therefore, bimaxillary osteotomy is a frequent surgery and potentially painful in adults. Bimaxillary surgery under general anesthesia is the common practice. And peripheral non-ultrasound-guided peripheral nerve blocks are widely used by surgeons. These minor blockades are used to avoid the undesired effects of anesthetics and analgesics; mainly the adverse respiratory effects of opioids. The practice of loco-regional anesthesia provides a control of perioperative pain in a multimodal way showing effective postoperative analgesia and minimizing the respiratory depression caused by the excess use of opioids.

In general, during bimaxillary surgery the surgeon performs the infiltrations with local anesthetic (LA) in a pre-incisional manner for the blockade of the terminal branches of the maxillary nerve intraorally and intranasally. The choice of LA is influenced by considerations such as the start of action, duration and toxicity. A wide range of LA has been used in maxillofacial surgery, such as lidocaine and ropivacaine among others. Both LA produce a reversible blockade of the sodium channel of the neuronal membrane, and are synthetic derivatives of cocaine. Both possess three essential functional units (hydrophilic tertiary amide chain, linked by an intermediate amide chain, to another lipophilic aromatic ring-portion). This means, both LA are amide type; but even if they belong to the same group of LAs there is still great differences in the beginning of action, duration of action and toxicity. Lidocaine has a faster start of action (short latency) than ropivacaine, and has an antiarrhythmic effect. Ropivacaine is more potent, the action last longer than lidocaine, and is less cardiotoxic than other equipotent LA such as bupivacaine and levobupivacaine.

Subsequently, the introduction of loco-regional nerve blocks has meant for the anesthesiologist, in the last three decades, a revolution in the management and control of perioperative pain. The expansion of the practice of loco-regional nerve blocks has been seen in both upper and lower limbs, as well as in trunk and abdomen. On the contrary, the facial blockages (both superficial and deep) have not experienced the same; laying its practice to the surgeon, or to anesthesiologists working on the chronic pain domain. The subsequent introduction of ultrasonography (USG) in the 1990s in the perioperative period also represented an important advance for anesthesiologist both in terms of safety and in terms of ease of management of venous and arterial catheterizations, and practice of loco-regional blockages. Consequently, USG experienced anesthesiologists have recently published in regards to the use of ultrasounds (US) for the blockage of facial nerves in children and adults undergoing maxillofacial surgery. USG devices are increasingly accessible, more portable, cheaper and safer; and therefore, its introduction in the field of perioperative pain management of maxillofacial surgery has still a long way to go.

The maxillary nerve, just like the ophthalmic, is only sensitive. It is detached from the anterolateral border of the trigeminal ganglion, laterally to the ophthalmic. From its origin, it goes above, crosses the foramen rotundum and penetrates into the background of the infratemporal fossa until it enters the pterygopalatine fossa (except the middle meningeal nerve, all its branches reach the pterygopalatine fossa before reaching the facies). In the pterygopalatine fossa the maxillary nerve is located in the upper part of the cavity and passes superiorly to the maxillary artery and superolaterally to the pterygopalatine ganglion. The maxillary nerve receives and conducts the sensitivity of the skin of the cheek, the lower eyelid, the wing of the nose and the upper lip. Its deep branches drive the sensitivity of the mucosa of the lower part of the nasal cavities or respiratory area, and of the dental roots and the gums of the maxilla.

Therefore, in order to produce an effective anesthesia of the maxillary area, the needle can be introduced through the pterygomaxillary fissure to the pterygopalatine fossa, with risk of vascular and nerve puncture. However, with real-time vision of the ultrasound-guided block, these risks will be limited, allowing a direct localization of the maxillary artery, position of the needle and the distribution of LA within the pterygopalatine fossa. The pterygopalatine fossa is anatomically deep and surrounded by bones. The most optimal ultrasound window is the infrazygomatic path, allowing the visualization of the entire axis of the pterygopalatine fossa up to the foramen rotundum.

The usual practice for the ultrasound-guided maxillary nerve block is the placement of the ultrasound probe in an infrazygomatic position and the introduction of the needle by suprazygomatic route for better visualization of the procedure. The approach by suprazygomatic route from the frontozygomatic angle is one of the safest and recommended routes to reach the foramen rotundum. This trajectory limits the insertion of the needle in the anterior portion of the foramen rotundum, avoiding, this way, the inadvertent puncture of the intraorbital content through the infraorbital fissure.

Experienced anesthesiologists in anesthesia for maxillofacial surgery, perform bilateral ultrasound-guided blockade of the maxillary nerve by suprazygomatic route with ropivacaine for greater control of perioperative pain. These investigators avoid the use of a combination of LA for maxillary nerve block. The combination of several local anesthetics in the same nerve block is sometimes used in perioperative anesthesia with the intention of compensating the short duration of action of some agents whose start of action is fast, such as lidocaine, and the high latency of the agents that present a more lasting action, such as ropivacaine. The combination of lidocaine and ropivacaine offers clinical advantages (rapid onset, long duration). However, to date, indications for combining LA are scarce because of the use of catheters in many forms of regional anesthesia that allow to prolong the duration of the block. This is nevertheless not an extended practice among anesthesiologists in maxillofacial surgery. On the other hand, it is important to also remember avoiding the use of maximum doses of two LA combined, which is based on the erroneous belief that their toxicities are independent; on the contrary, the toxicities have an additive character.

Multiple drugs have been used to increase the time of action of LA, such as adrenaline, clonidine, dexamethasone, ketamine and dexmedetomidine, among others. To the study patients, adrenaline is always administered along with physiological serum by the surgeon at the local level to improve the surgical field, both in patients who undergo pre-incision infiltration and bilateral blockade of the maxillary nerve. The use of Clonidine is ruled out because it is not supplied in the hospital center where the investigators will carry out the study. The use of dexamethasone and ketamine is ruled out, because they will be administered intravenously in the patient's perioperative period as anti-inflammatory agents and anesthetic adjuvant, respectively. And the use of Dexmedetomidine is also ruled out in order to prolong the effect of the nerve blockade as this indication is not in the technical file.

ELIGIBILITY:
Inclusion Criteria:

* patients who undergo scheduled bimaxillary surgery

Exclusion Criteria:

* the refusal to participate in the study,
* patients who are scheduled for bimaxillary surgery together with another complementary surgical procedure (such as mentoplasty, rhinoplasty, blepharoplasty),
* age <18 years,
* reinterventions,
* urgent surgeries,
* allergies to local anesthetics,
* allergies to anti-inflammatories agents,
* allergies to opioids,
* American Society of Anesthesiologists Physical Status Classification (ASA) ≥3

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Opioids consumption | 2hours postoperatively
  evaluation of the effectiveness of the bilateral ultrasound-guided blockade with ropivacaine by suprazygomatic route, compared to the peripheral infiltration of the nerve with lidocaine and adrenaline, on the consumption of opioids for control of perioperative pain of patients intervened of elective bimaxillary osteotomy, evaluated by means of the analogical visual scale of pain in the immediate postoperative period (2 hours postoperatively).
comparison of the use of opioids in the intraoperative period | intraoperatively
  comparison of the use of opioids in the intraoperative period (Target Controlled Infusion (TCI) ng / ml - intravenous remifentanil),

SECONDARY OUTCOMES:
comparison of the use of rescue opioids in the postoperative period in hospitalization | (2-18hours postoperative)
  comparison of the use of rescue opioids (milligrams of intravenous methadone) in the postoperative period in hospitalization (2-18hours postoperative)
the comparison of the incidence of immediate postoperative nausea and vomiting (PONV) | 0-18hours after surgery
  the comparison of the incidence of immediate postoperative nausea and vomiting (PONV) in resuscitation and up to 18 hours after surgery
registry of complications derived from ultrasound-guided maxillary nerve block. | 0-18hours after surgery
  registry of complications derived from ultrasound-guided maxillary nerve block.

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Molins, Principal Investigator — Anesthesiologist- Anestalia
Locations (1):
- Centro Medico Teknon - Grupo Quirón Salud, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of the study completion
Access Criteria: data access requests will be reviewed by an external independent Review Panel. Requestors will be required to sign a Data Access Agreement

REFERENCES:
- [Derived] Molins G, Valls-Ontanon A, De Nadal M, Hernandez-Alfaro F. Ultrasound-Guided Suprazygomatic Maxillary Nerve Block Is Effective in Reducing Postoperative Opioid Use Following Bimaxillary Osteotomy. J Oral Maxillofac Surg. 2024 Apr;82(4):412-421. doi: 10.1016/j.joms.2023.12.018. Epub 2024 Jan 2. PMID 38253318

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/29/NCT03913429/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/29/NCT03913429/ICF_001.pdf